CLINICAL TRIAL: NCT02510703
Title: Assessment of Coronary Endothelial Function in Diabetic Patients With Acute Coronary Syndrome Using 15O-water Positron Emission Tomography
Acronym: D-TEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-085
Record Dates: First submitted 2015-07-27; First posted 2015-07-29 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2015-08

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Type 2 diabetes group (Other): Type 2 diabetes group
  Interventions: Other: Coronary endothelial function measurements by quantitative method (TEP at 15O-H2O)
- no diabetes (Other): no diabetes
  Interventions: Other: Coronary endothelial function measurements by quantitative method (TEP at 15O-H2O)

INTERVENTIONS:
Other: Coronary endothelial function measurements by quantitative method (TEP at 15O-H2O)

SUMMARY:
Type 2 diabetes is associated with early and diffuse abnormalities of endothelial function, especially in the coronary arteries, which are a factor of poor prognosis. Following acute coronary syndrome, the endothelial function abnormalities usually persist for several weeks before regressing. Their persistence 6-8 weeks after myocardial infarction is a poor prognostic factor. Investigators assume that global abnormalities of endothelial function in patients with diabetes may be additive with segmental abnormalities in revascularized myocardium, and contribute to worsening the prognosis in these patients. Furthermore, there is no published data showing any relationship between calcium score and endothelial function abnormalities in these patients. The investigators seek a relationship between calcium score and persistence of abnormalities of coronary endothelial function in these patients.

The main objective of this study was to compare coronary endothelial function by quantitative method (TEP at 15O-H2O) in diabetic patients and nondiabetic following acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a first myocardial infarction, type 2 diabetic or non-diabetic treated by angioplasty in acute phase (TIMI 3)
* Myocardial viability test before discharge
* Age over 18 years
* Informed Consent dated and signed by the patient
* Written and spoken French
* Beneficiary of social security insurance

Exclusion Criteria:

* Hypertension> 160/90 mmHg despite medical treatment
* Lack of effective revascularization in acute phase of myocardial infarction (TIMI grade <3)
* Significant three-vessel coronary artery disease (> 70% stenosis in the other two coronary arteries); occlusion of a coronary artery; schedule revascularization (percutaneous or surgical); left main coronary artery stenosis
* Previous history of myocardial infarction
* Mechanical complication (mitral regurgitation, ventricular septal rupture, left ventricular free wall rupture)
* Heart failure
* No myocardial viability test before discharge, for whatever reason
* Type 1 diabetes
* Pregnant and / or lactating
* Age under 18 years or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Comparison of quantitative variables coronary endothelial function in PET according to the presence or absence of type 2 diabetes in patients investigated with the waning of a first heart attack | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Cardiologie, Caen, France